CLINICAL TRIAL: NCT01566110
Title: A Randomized Controlled Trial to Evaluate the Efficacy and Safety of a Gluten-Free Diet in Patients With Asymptomatic Celiac Disease and Type 1 Diabetes, Celiac Disease and Diabetes - Dietary Intervention and Evaluation Trial (CD-DIET)
Brief Title: Celiac Disease and Diabetes- Dietary Intervention and Evaluation Trial
Acronym: CD-DIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Farid Mahmud, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000030346
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Celiac Disease; Diabetes Mellitus, Type 1
Keywords: pediatric; dietary treatment; celiac disease; T1D
MeSH Terms: conditions — Celiac Disease; Diabetes Mellitus, Type 1 | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet Intervention Group (Experimental)
  Interventions: Dietary Supplement: Gluten Free Diet
- Control Group (No Intervention): Subjects assigned to the control group will continue their usual diet. They will receive dietary teaching at each study visit as part of their diabetes management.

INTERVENTIONS:
Dietary Supplement: Gluten Free Diet — Subjects assigned to the intervention group will receive a standardized dietary education intervention that will inform subjects and family members of the effects of gluten on the gastrointestinal tract and emphasize the need to adhere to a diet that is gluten-free. This intervention will be delivered by a dietician who is trained in celiac disease and gluten free diet.
  Arms: Diet Intervention Group

SUMMARY:
Currently no consensus exists on the optimal way to manage asymptomatic patients with celiac disease (CD) and Type 1 diabetes (T1D). The impact of dietary treatment as it pertains to clinically relevant outcomes such as metabolic control, bone mineralization and wellbeing will be evaluated in this study. A randomized controlled study longitudinally evaluating HbA1c and glycemic excursions using continuous glucose monitoring will rigorously determine the impact of a gluten-free diet (GFD) on blood glucose variability in patients with T1D.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet each of the following criteria for inclusion into the study:

1. Males and females age between 8 and 45 years.
2. Diagnosis of T1D by American Diabetes Association (ADA) criteria with duration of T1D greater than 1 year.
3. CD screen positive (Positive TTG serology).
4. Presence of a positive duodenal biopsy for CD (Marsh score of 2 or greater).
5. Ability of the subject or a legally authorized representative to speak and read English or French.
6. Ability of the subject to participate in all aspects of this clinical trial.
7. Written informed consent must be obtained and documented, with assent of the child if <14 years of age.

Exclusion Criteria:

1. Prior diagnosis of CD.
2. Symptoms or other evidence of overt CD defined by at least one of:

   * CD symptoms using the Gastrointestinal Symptom Scale [GISS]
   * Impaired growth
   * Anemia
3. Presence of recurrent apthous ulcers (painful mouth ulcers involving mucous membranes) or dermatitis herpetiformis (blistering skin rash). Mouth or skin lesions known to be related to diagnosed herpes are not included in this exclusion criteria.
4. Conditions which in the opinion of the investigator may interfere with the subject's ability to participate in the study.
5. Prior enrolment in the current study.
6. Concurrent enrolment in a longitudinal intervention study.
7. Previously diagnosed or treated osteoporosis.
8. Pregnancy or lactation.

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Metabolic Control | Change from Baseline over 1 year
  As a standard measure of diabetes control, HbA1c is assessed on a frequent and regular basis as recommended by the CDA 2008 guidelines in both pediatric and adult patients. HbA1c is synthesized throughout the cycle of a red blood cell and reflects the degree of chronic hyperglycemia present in patients with diabetes.

SECONDARY OUTCOMES:
Hypoglycemic Episodes | Frequency over 12 months
  The frequency and severity of hypoglycemic episodes will be recorded at each clinic visit. These will be classified as severe hypoglycemic episodes in subjects with normal hypoglycemic awareness.
Continuous Glucose Monitoring | Baseline, 6 months and 12 months after randomization
  Data will be evaluated for data quality, overall mean glucose, overall variability of blood glucose, patterns of blood glucose excursion, and measures of quality of glycemic control.

CONTACTS AND LOCATIONS:
Overall Officials: Farid Mahmud, MD, Principal Investigator — The Hospital for Sick Children
Locations (7):
- Canada (7):
  - McMaster University, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences, London, Ontario
  - St. Joseph's Healthcare, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - LMC Diabetes and Endocrinology, Toronto, Ontario

REFERENCES:
- [Derived] De Melo EN, Clarke ABM, McDonald C, Saibil F, Lochnan HA, Punthakee Z, Assor E, Marcon MA, Mahmud FH. Gastrointestinal Symptoms in Type 1 Diabetes: Relationship With Autoimmune and Microvascular Complications. J Clin Endocrinol Metab. 2022 May 17;107(6):e2431-e2437. doi: 10.1210/clinem/dgac093. PMID 35176765
- [Derived] Gould MJ, Mahmud FH, Clarke ABM, McDonald C, Saibil F, Punthakee Z, Marcon MA. Accuracy of Screening Tests for Celiac Disease in Asymptomatic Patients With Type 1 Diabetes. Am J Gastroenterol. 2021 Jul 1;116(7):1545-1549. doi: 10.14309/ajg.0000000000001193. PMID 33852450
- [Derived] Weiman DI, Mahmud FH, Clarke ABM, Assor E, McDonald C, Saibil F, Lochnan HA, Punthakee Z, Marcon MA; CD-DIET Study Group. Impact of a Gluten-Free Diet on Quality of Life and Health Perception in Patients With Type 1 Diabetes and Asymptomatic Celiac Disease. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e1984-e1992. doi: 10.1210/clinem/dgaa977. PMID 33524131
- [Derived] Mahmud FH, Clarke ABM, Joachim KC, Assor E, McDonald C, Saibil F, Lochnan HA, Punthakee Z, Parikh A, Advani A, Shah BR, Perkins BA, Zuijdwijk CS, Mack DR, Koltin D, De Melo EN, Hsieh E, Mukerji G, Gilbert J, Bax K, Lawson ML, Cino M, Beaton MD, Saloojee NA, Lou O, Gallego PH, Bercik P, Houlden RL, Aronson R, Kirsch SE, Paterson WG, Marcon MA. Screening and Treatment Outcomes in Adults and Children With Type 1 Diabetes and Asymptomatic Celiac Disease: The CD-DIET Study. Diabetes Care. 2020 Jul;43(7):1553-1556. doi: 10.2337/dc19-1944. Epub 2020 Apr 28. PMID 32345653
- [Derived] Assor E, Marcon MA, Hamilton N, Fry M, Cooper T, Mahmud FH. Design of a dietary intervention to assess the impact of a gluten-free diet in a population with type 1 Diabetes and Celiac Disease. BMC Gastroenterol. 2015 Dec 21;15:181. doi: 10.1186/s12876-015-0413-0. PMID 26692164
- [Derived] Mahmud FH, De Melo EN, Noordin K, Assor E, Sahota K, Davies-Shaw J, Cutz E, Somers G, Lawson M, Mack DR, Gallego P, McDonald C, Beaton MD, Bax K, Saibil F, Gilbert J, Kirsch S, Perkins BA, Cino M, Szentgyorgyi E, Koltin D, Parikh A, Mukerji G, Advani A, Lou O, Marcon MA. The Celiac Disease and Diabetes-Dietary Intervention and Evaluation Trial (CD-DIET) protocol: a randomised controlled study to evaluate treatment of asymptomatic coeliac disease in type 1 diabetes. BMJ Open. 2015 May 11;5(5):e008097. doi: 10.1136/bmjopen-2015-008097. PMID 25968008